CLINICAL TRIAL: NCT04328909
Title: Pilot Trial of a Software Application to Facilitate Communication and Shared Decision-making With Parents of Febrile Infants
Brief Title: Study of an App to Facilitate Communication With Parents of Febrile Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2000027687; 1K08HS026006-01A1 (AHRQ)
Record Dates: First submitted 2020-03-19; First posted 2020-04-01 (Actual); Last update posted 2022-02-03 (Actual); Status verified 2022-02

CONDITIONS: Fever
MeSH Terms: conditions — Fever | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- E-Care (Experimental): Parent-centered care software application (e-Care) to ensure parents of febrile infants are optimally informed and participate in shared decision making in the ED
  Interventions: Device: E-Care
- Control Group (Active Comparator): Usual care - No E-Care app will be provided
  Interventions: Other: Control Group

INTERVENTIONS:
Device: E-Care — Parent-centered care software application (e-Care) to ensure parents of febrile infants are optimally informed and participate in shared decision making in the ED
  Arms: E-Care
Other: Control Group — Usual care - No E-Care app will be provided
  Arms: Control Group

SUMMARY:
The objective of this research project is to test an evidence-based parent-centered care software application (e-Care) to ensure that parents of febrile infants from a wide range of socio-demographic backgrounds are optimally informed despite being fatigued and stressed, and able to participate in shared decision making (SDM) in the unfamiliar, time-pressured environment of the Emergency Department (ED)

DETAILED DESCRIPTION:
Recruitment and Consent: Pediatric emergency medicine fellows and attending physicians will be enrolled at a Section meeting or individually and not during patient care in the ED. Written informed consent will be obtained. For physicians who decline enrollment, parents of febrile infants will not be approached for enrollment. Each pediatric emergency medicine fellow and attending physician will be assigned a unique study identifier.

Parents will be enrolled in the Yale New Haven Children's Hospital pediatric ED. The RA or PI will be notified by the triage nurse, bedside nurse, or treating pediatric emergency medicine fellow or attending physician of an eligible parent of a febrile infant, defined as an infant with a documented temperature of ≥38.0° C (100.4° F) in the ED or within the past 24 hours at home or in clinic who is evaluated in the pediatric ED at Yale New Haven Children's Hospital. After introduction by the treating medical team, the RA or PI will approach eligible parent(s) for enrollment when they are in the ED examination room and after initial discussion with the pediatric emergency medicine fellow or attending physician. Study procedures and the risks/benefits of participating will be described, and written informed consent will be obtained. When more than one parent is available, the parents will be asked to identify who will complete all study forms.

All parents will receive a unique study identifier. This unique study identifier will be linked to the signed informed consent document and to the infant's MRN. The infant's MRN will be recorded on an excel file stored on the Yale ITS managed, encrypted, password-protected laptop that is stored in the PI's locked office.

Baseline (Month 1): Parents will complete a baseline demographics form (please see Data Collection below) and will complete an outcome measures survey at the time of disposition from the ED and 1 week after the ED visit

Intervention (e-Care) Group: After enrollment of a parent, the RA or PI will provide a brief orientation of e-Care to the treating pediatric emergency medicine fellow and/or attending physician, including showing the "What happens after the test results are known" section for parents of infants 29-60 days of age. The parent will complete a baseline demographics form.The e-Care app will then be provided to the parent on an iPad with a brief overview of the app provided by the RA or PI. The parent will then view the e-Care app at his or her discretion throughout the duration of the ED visit. At the time of disposition from the ED, parents will complete an outcome measures survey and an acceptability survey, and 1 week after the ED visit, parents will complete another outcome measures survey. Parents will also answer brief qualitative questions at the time of disposition.The RA or PI will extract de-identified data on the infant from the Epic electronic health record and will confirm some of the data on a phone call with parents 1 week after the ED visit. Physicians will complete an acceptability survey and answer brief qualitative questions at the time of the infant's disposition from the ED.

Control Group: For parents/febrile infant dyads who are randomized to usual care, no e-Care app will be provided. Outcome measures will be completed as described for the Intervention group, with the exception that no acceptability surveys or qualitative questions will be completed by parents and no acceptability survey will be completed by physicians.

ELIGIBILITY:
Inclusion Criteria for Parents - Parents of febrile infants ≤60 days of age (fever defined as a documented temperature of ≥38.0° C (100.4° F) in the ED or within the past 24 hours at home or in clinic)

Exclusion Criteria for Parents -

* Not comfortable with conversational and written English or Spanish
* Infant is critically ill and requiring life-saving interventions on arrival to the ED (e.g., endotracheal intubation, CPR)
* Parent has been previously enrolled

Inclusion Criteria for Physicians -

- Pediatric emergency medicine fellows and attending physicians from Yale School of Medicine (Section of Pediatric Emergency Medicine)

Exclusion Criteria for Physicians - none

Ages: 1 Day to 60 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2020-06-08 (Actual); Primary Completion 2021-07-28 (Actual); Study Completion 2021-08-09 (Actual)

PRIMARY OUTCOMES:
COMRADE scale | Administered at the end of the emergency department visit (4 hours after delivery of the intervention)
  This is a 20 statements survey (5-point Likert scale, Strongly Disagree to Strongly Agree). It is scored from 20 to 100. Higher scores indicate better respondent (parent) perceptions of risk communication and their confidence in the decision. Administration time is 2-3 minutes. This will be measured in both parents of infants <= 28 days and parents of infants 29 to 60 days.

SECONDARY OUTCOMES:
Knowledge questionnaire | Administered at the end of the emergency department visit (4 hours after delivery of the intervention)
  8 statements (True, False, Unsure), scored as a proportion of correct responses (minimum 0, maximum 8). Higher proportion of correct responses = higher knowledge. Administration time is 1-2 minutes.This will be measured in both parents of infants <= 28 days and parents of infants 29 to 60 days.
Anxiety Questionnaire | Administered at the end of the emergency department visit (4 hours after delivery of the intervention)
  This is a six-item version of the State-Trait Anxiety Inventory. There are 6 statements about how the parent feels at that moment (4-point Likert scale, rated from "Not at all" to "Very much so"). Scored from 6 to 24, with higher scores indicating higher anxiety. Administration time is 1 minute. This will be measured in both parents of infants <= 28 days and parents of infants 29 to 60 days.
Anxiety Questionnaire | Administered 1 week after emergency department visit
  This is a six-item version of the State-Trait Anxiety Inventory. There are 6 statements about how the parent feels at that moment (4-point Likert scale, rated from "Not at all" to "Very much so"). Scored from 6 to 24, with higher scores indicating higher anxiety. Administration time is 1 minute. This will be measured in both parents of infants <= 28 days and parents of infants 29 to 60 days.
Acceptability of e-Care for parents of infants <= 28 days | Administered at the end of the emergency department visit (4 hours after delivery of the intervention)
  One question with 3 statements asking parents how information was presented in the app (4-point scale, rated as "Poor" to "Excellent"), scored from 3 to 12 with higher scores=greater acceptability; Two questions asking about the length of the app and the amount of information presented (3-point scale, "Too short," "Too long," "Just right"); two questions asking ease of use and how helpful the app was (4-point scales); 2 open-ended questions; higher scores indicate greater acceptability. Administration time is 2-3 minutes.
Acceptability of e-Care for parents of infants 29 to 60 days | Administered at the end of the emergency department visit (4 hours after delivery of the intervention)
  One question with 4 statements asking parents how information was presented in the app (4-point scale, rated as "Poor" to "Excellent"), scored from 4 to 16 with higher scores=greater acceptability; Two questions asking about the length of the app and the amount of information presented (3-point scale, "Too short," "Too long," "Just right"); one question asking about balance in presentation of options (3-point scale); three questions asking ease of use and how helpful the app was (4-point scales); 2 open-ended questions; higher scores indicate greater acceptability. Administration time is 2-3 minutes.
Acceptability of E-Care for physicians | Administered at the end of the emergency department visit (4 hours after delivery of the intervention)
  10 statements (5-point Likert scale, Strongly Disagree to Strongly Agree). Scored from 10 to 50, with higher scores = greater acceptability. Administration time is 1-2 minutes.
Decision Regret scale | Administered 1 week after emergency department visit
  This is a 5 statements 5-point Likert scale, Strongly Disagree to Strongly Agree. Scored from 0 (no regret) to 100 (high regret). This will be measured in parents of infants 29 to 60 days
Decisional conflict scale | Administered at the end of the emergency department visit (4 hours after delivery of the intervention)
  This is a 10 statements (Yes, Unsure, No). Scored from 0 (no decisional conflict) to 100 (extremely high decisional conflict).This will only be measured for the parents of infants 29 to 60 days.
Values questionnaire | Administered at the end of the emergency department visit (4 hours after delivery of the intervention)
  This is a 2 questions with 2 statements each, whereby parents choose which of the 2 statements are more important to them (no score). Administration time 1 minute. This will be measured in the parents of infants 29 to 60 days
Verbal question for parents of infants <= 28 days | Administered at the end of the emergency department visit (4 hours after delivery of the intervention)
  Qualitative verbal question whether they viewed the app. This will be measured qualitatively (no score).
Verbal questions for parents of infants 29 to 60 days | Administered at the end of the emergency department visit (4 hours after delivery of the intervention)
  Qualitative verbal question whether they viewed the app and whether physicians showed them information in the app (intervention group only). This will be measured qualitatively (no score).
Verbal questions for parents for physicians | Administered at the end of the emergency department visit (4 hours after delivery of the intervention)
  about the app (if caring for parent in the intervention group) and question about how they communicated to parents (both groups). This will be measured qualitatively (no score).

CONTACTS AND LOCATIONS:
Locations (1):
- Yale New Haven Hospital, New Haven, Connecticut, United States